CLINICAL TRIAL: NCT06073080
Title: Recovery Protein Nutrition as a Countermeasure for Anabolic Resistance Following Sleep Loss
Acronym: PSL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-27H
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sleep, Inadequate
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Randomized, parallel arm study. All volunteers will complete a sleep satiated phase and sleep restriction phase before randomized allocation to either an even protein nutrition intervention or a skewed protein nutrition intervention during a recovery phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Nutrition Even (Experimental): Volunteers will consume 1.6 g protein/kg/d as an even (~0.4/0.4/0.4/0.4 g/kg) distribution across breakfast, lunch, dinner, and a snack.
  Interventions: Other: Protein Nutrition During Recovery
- Protein Nutrition Skewed (Active Comparator): Volunteers will consume 1.6 g protein/kg/d as a skewed (~0.11/0.27/1.15/0.07 g/kg) distribution across breakfast, lunch, dinner, and a snack.
  Interventions: Other: Protein Nutrition During Recovery

INTERVENTIONS:
Other: Protein Nutrition During Recovery — Dietary Protein Nutrition Distribution

SUMMARY:
The current study will determine protein nutritional status (MPS and WBPB) in response to military-relevant sleep loss, and whether an even protein nutrition distribution during recovery optimally supports MPS and WBPB. Adults (n=20) will complete a 7d sleep satiated phase (~7-9h target/d), a 4d military-relevant sleep restriction phase (~4h /d), and a 3d recovery phase (~7-9h target/d) in a randomized, parallel design. During recovery, volunteers will consume 1.6 g protein/kg/d as an even (~0.4/0.4/0.4/0.4 g/kg) or skewed (~0.11/0.27/1.15/0.07 g/kg) distribution. Sleep will be monitored throughout the study using wrist actigraphy and diaries. During each phase, integrated daily MPS will be estimated using ingested deuterium oxide, salivary and blood sampling, and muscle biopsies, while WBPB will be estimated using ingested 15-N alanine and urine collections. At the end of each phase, metabolic testing will be used to assess the effects of sleep loss on substrate utilization and include consuming a carbohydrate beverage, serial blood draws, indirect calorimetry, and steady-state aerobic exercise. The knowledge products derived from the proposed effort will be informative to next generation ration development and support military-specific recovery nutrition guidance following operations involving sleep loss.

DETAILED DESCRIPTION:
The nutritional fitness of Service Members directly influences recovery from operational stress. Inadequate recovery nutrition following military missions, including sleep loss, exacerbates skeletal muscle loss and contributes to degraded physical performance. Muscle loss and performance declines following stress are in part due to inadequate nutritional fitness, impaired muscle recovery, and negative whole-body protein balance (WBPB). Sleep loss dysregulates anabolic hormones, induces catabolism, and reduces muscle protein synthesis (MPS). However, WBPB has not been assessed following military-relevant sleep loss (i.e., 4h/d) alone. This presents an important knowledge gap given the influence of WBPB on health and readiness. Consuming increased dietary protein following sleep loss could enhance muscle recovery by stimulating MPS and supporting WBPB, but whether protein recovery nutrition counteracts the stress of sleep loss is unknown. Beyond the quantity of protein consumed, optimizing the timing/distribution of daily protein consumption is required to augment anabolism. Consuming a skewed protein distribution results in meals (i.e., breakfast and lunch) that deliver a suboptimal protein quantity for maximally stimulating MPS. Alternatively, targeting an even protein distribution may optimize anabolism and recovery following stress by providing per meal protein quantities that maximally stimulate MPS and support WBPB. The efficacy of manipulating protein distribution for counteracting the stress of sleep loss is unknown. The proposed effort will determine protein nutritional status (MPS and WBPB) in response to military-relevant sleep loss, and whether an even protein nutrition distribution during recovery optimally supports MPS and WBPB. Adults (n=20) will complete a 7d sleep satiated phase (~7-9h target/d), a 4d military-relevant sleep restriction phase (~4h /d), and a 3d recovery phase (~7-9h target/d) in a randomized, parallel design. During recovery, volunteers will consume 1.6 g protein/kg/d as an even (~0.4/0.4/0.4/0.4 g/kg) or skewed (~0.11/0.27/1.15/0.07 g/kg) distribution. Sleep will be monitored throughout the study using wrist actigraphy and diaries. During each phase, integrated daily MPS will be estimated using ingested deuterium oxide, salivary and blood sampling, and muscle biopsies, while WBPB will be estimated using ingested 15-N alanine and urine collections. At the end of each phase, metabolic testing will be used to assess the effects of sleep loss on substrate utilization and include consuming a carbohydrate beverage, serial blood draws, indirect calorimetry, and steady-state aerobic exercise. The knowledge products derived from the proposed effort will be informative to next generation ration development and support military-specific recovery nutrition guidance following operations involving sleep loss.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 - 39 years
* Body mass index < 30.0 kg/m2
* Self-report weight stable for the past 2 months (± ~3 kg)
* Healthy without evidence of chronic illness, musculoskeletal injury, or diagnosed sleep disorder (i.e., insomnia) as determined by the USARIEM Office of Medical Support and Oversight (OMSO) or home duty station medical support
* Self-report participates in aerobic and/or resistance exercise, on average, ≥2 days per week for previous 6 months
* Willing to refrain from alcohol, smoking/using any nicotine product (includes e-cigarettes, vaping, chewing tobacco), caffeine, and dietary supplements during the intervention periods of the study
* Supervisor approval for federal civilian employees and non-HRV active duty military personnel
* Biological females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or able to provide self-report documentation of sustained (i.e., ~ >3 months) oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous hormonal levels (i.e., IUD or no oral placebos)

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., abnormal blood clotting, kidney disease, diabetes, cardiovascular disease, anemia etc.) as determined by OMSO or home duty station medical support
* History of complications with lidocaine (or similar local anesthetic)
* Present condition of substance abuse (e.g., alcoholism, anabolic steroid use etc.) as self-report or determined by OMSO or home duty station medical support
* Cumulative blood donation of greater than 550mL within 8-wk of beginning scheduled study blood collection
* Cumulative blood donation of greater than 550mL within 8-wk after completing scheduled study blood collection
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test prior to body composition scans and self-report for breastfeeding)
* Unwilling or unable to consume study diets or foods provided due to personal preference, dietary restrictions, and/or food allergies
* Unwilling or unable to adhere to study physical restrictions or sleep prescriptions

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Whole-body Protein Balance | 24 hours
  15N labeled stable isotope
Integrated Muscle Protein Synthesis | 72 hours
  deuterium oxide integrated stable isotope

CONTACTS AND LOCATIONS:
Overall Officials: Jess A Gwin, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

DOCUMENTS (1):
  • Informed Consent Form (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT06073080/ICF_000.pdf